CLINICAL TRIAL: NCT04248400
Title: Effectiveness of Tai Chi to Improve Cognitive Function in Older Adults With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Tai Chi to Improve Cognitive Function in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCMCI
Record Dates: First submitted 2020-01-16; First posted 2020-01-30 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Conventional exercise (Active Comparator): A 24 weeks conventional exercise training with three 1-hour section per week
  Interventions: Other: Conventional exercise
- Tai Chi (Experimental): A 24 weeks Tai Chi training with three 1-hour section per week
  Interventions: Other: Tai Chi training

INTERVENTIONS:
Other: Tai Chi training — A 24 weeks Tai Chi training with three 1-hour section per week
  Arms: Tai Chi
Other: Conventional exercise — A 24 weeks conventional exercise training with three 1-hour section per week
  Arms: Conventional exercise

SUMMARY:
Mild cognitive impairment (MCI) is a transitional state between normal cognitive decline and dementia. Individuals with MCI are having an impairment in cognitive function compared with normal age-matched counterparts, while their cognitive function is still sufficient for their daily function. The prevalent rate of MCI is ranging from 10% to 20%. Patients with MCI are more susceptible to dementia with annual conversion rate between 5% and 20%. It is well-known that dementia not only lead to devastating consequences to the patients and their care-givers, but also immense healthcare and socioeconomic burdens. The growing prevalence of MCI in our rapidly aging population warrants immediate action to identify effective interventions to prevent progression of the cognitive impairment and its conversion to dementia. Currently, there is no pharmaceutical treatment proven to be effective in alleviating the cognitive decline in MCI patients. Nonetheless, previous researches have demonstrated that mind activity, physical exercise and social engagement are all have positive effects in alleviating the cognitive decline in MCI patients. Tai Chi is a traditional form of Chinese mind-body exercise that consists of both physical exercise and meditation component. Practicing Tai Chi can also facilitate social engagement as people usually practice in group. Tai Chi is expected to be more acceptable to the older adults for incorporating it with their daily life to preserve cognitive function, compared with conventional physical activity modalities (e.g., running/jogging and gym-based resistance training). Preliminary evidences suggest the potential of Tai Chi for alleviating cognitive decline in older adults.

A randomized controlled trial is needed to conclude on the therapeutic use of Tai Chi before it can be large-scale implemented at community level. This study seeks to extend previous findings of the beneficial effects of Tai Chi on cognitive function in older adults with MCI and examine the impact of Tai Chi training in protecting older adults with MCI from developing dementia. This study also attempt to delineate the behind mechanism of Tai Chi on alleviating cognitive decline by including measurements in neuroimaging and blood markers.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged equal or larger than 50 years
* Ethnic Chinese
* MCI under criteria of Mayo Clinic, including the following:

  i. Participants have noticed a decline in their cognitive function ii. The total score of participants in age and education corrected Hong Kong version Montreal Cognitive assessment is below the 7th percentile of the normative data from Hong Kong iii. The decline of cognitive function does not affect the daily function of the participants revealed by getting ≥2 marks in every item of Chinese Lawton Instrumental Activities of Daily Living Scale (4-point Scale)

Exclusion Criteria:

* History of major diseases such as cancer, stroke, cardio-/cerebrovascular, neurodegenerative and renal diseases,
* Diagnosis of dementia or using anti-dementia medication,
* Diagnosis of psychiatric disease or using psychiatric medication,
* Inability to perform exercise,
* Regular mind-body exercise habit (>3 times 60-minute Tai Chi, yoga or Qigong weekly),
* Physically active (>150 minutes of moderate-intensity physical activity or >75 minutes of vigorous-intensity physical activity weekly)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The score of the Montreal Cognitive Assessment | 12 weeks
  Change in the score of the Montreal Cognitive Assessment. The score ranged from 0 to 30. Higher score indicates a better cognitive function
The score of the Montreal Cognitive Assessment | 24 weeks
  Change in the score of the Montreal Cognitive Assessment. The score ranged from 0 to 30. Higher score indicates a better cognitive function

SECONDARY OUTCOMES:
30-min delay recall | 12 weeks and 24 weeks
  The 30-min delay recall test assesses long term memory. Ten words will be read to the participants. The participants will have to recall the 10 words after 30 minutes.
Trial making test | 12 weeks and 24 weeks
  Executive function will be trial making test. The participants will be asked to connect a number of dots according to particular sequence. The time needed for the participant to connect all dots will be recorded. The shorter time the participant needed to connect all dots correctly indicate the better executive function of the participant
Stroop test | 12 weeks and 24 weeks
  Attention will be assessed by stroop test. During the test, participants need to read out the colour of dots or words. The time needed to correctly named all colour of dots/words will be recorded. The faster the participant finished the test indicate the better attention of the participant
Verbal fluency | 12 weeks and 24 weeks
  Verbal fluency test assesses the language domain of cognitive function. Participants need to name animals/ vegetable/ fruits as much as positive in 1 minutes. The more the participant named, the better of their language ability
Digit span | 12 weeks and 24 weeks
  Working Memory will be assessed by digit span. Digit Span Forward requires the participants to repeat numbers in the same order as read by the assessors, and Digit Span Backward requires the participants to repeat the numbers in the reverse order of that presented by the assessors.
n-back test | 12 weeks and 24 weeks
  Short term memory will be assessed by n-back test.

CONTACTS AND LOCATIONS:
Overall Officials: Parco Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu AP, Chin EC, Yu DJ, Fong DY, Cheng CP, Hu X, Wei GX, Siu PM. Tai Chi versus conventional exercise for improving cognitive function in older adults: a pilot randomized controlled trial. Sci Rep. 2022 May 25;12(1):8868. doi: 10.1038/s41598-022-12526-5. PMID 35614144